CLINICAL TRIAL: NCT00845195
Title: Comparison of Seasonal Allergic Rhinitis Treatment With 2 Antihistamines Used in Combination With Intranasal Corticosteroid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Michael Edwards, PhD\Global Medical Affairs- Allergy, Alcon Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMA-08-23
Record Dates: First submitted 2009-02-13; First posted 2009-02-18 (Estimated); Results first posted 2010-04-21 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: Rhinitis; Allergy; Nasal Spray; Antihistamine; Intranasal Corticosteroid
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olopatadine HCl Nasal Spray, 0.6% (Experimental)
  Interventions: Drug: Olopatadine HCl Nasal Spray, 0.6%
- Azelastine HCl Nasal Spray, 0.1% (Active Comparator)
  Interventions: Drug: Azelastine HCl Nasal Spray, 0.1%

INTERVENTIONS:
Drug: Olopatadine HCl Nasal Spray, 0.6% — 2 sprays/nostril, twice daily (in addition to Fluticasone Propionate Nasal Spray 50 mcg 2 sprays/nostril once daily) for 14 +/- 3 days
  Arms: Olopatadine HCl Nasal Spray, 0.6%
Drug: Azelastine HCl Nasal Spray, 0.1% — 2 sprays/nostril, twice daily (in addition to Fluticasone Propionate Nasal Spray 50 mcg 2 sprays/nostril once daily) for 14 +/- 3 days
  Arms: Azelastine HCl Nasal Spray, 0.1%

SUMMARY:
The purpose of this study is to compare the efficacy of Olopatadine Nasal Spray with Azelastine Nasal Spray when treatments are utilized in conjunction with Fluticasone Nasal Spray for the treatment of seasonal allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide consent/assent
* History of spring/summer allergic rhinitis
* Positive skin prick and/or intradermal test
* Absence of significant anatomic abnormalities, infection, bleeding, and mucosal ulcerations
* Non-pregnant (where applicable)
* Able to complete daily diary

Exclusion Criteria:

* Smoker
* Concurrent disease such as rhinitis medicamentosa or large obstructive nasal polyps
* History of current chronic sinusitis
* Asthma
* Use of anti-allergy immunotherapy, corticosteroids, chronic use of long acting antihistamines
* History of severe, unstable, or uncontrolled cardiovascular, hepatic, renal and/or other diseases/illnesses
* History or evidence of nasolacrimal drainage system malfunction

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center for Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 8, 2009 - April 22, 2009
Groups:
- Olopatadine HCl Nasal Spray, 0.6%: Olopatadine HCL Nasal Spray, 0.6% + Fluticasone Propionate Spray, 50 mcg
- Azelastine HCl Nasal Spray, 0.1%: Azelastine HCL Nasal Spray, 137 mcg + Fluticasone Propionate Spray, 50 mcg
Period: Overall Study
Arm/Group | Olopatadine HCl Nasal Spray, 0.6% | Azelastine HCl Nasal Spray, 0.1%
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olopatadine HCl Nasal Spray, 0.6% | Azelastine HCl Nasal Spray, 0.1% | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 69 | 70 | 139
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 45 | 81
  Male | 39 | 30 | 69

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Reflective Total Nasal Symptom Score (rTNSS) From Baseline
Description: Responses to patient-completed diaries for reflective Total Nasal Symptom Scores (rTNSS). TNSS is composed of 4 individual assessments, which included runny nose, itchy nose, stuffy nose, and sneezing; each of the 4 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 4 assessments are then added together for a composite score (TNSS score), the maximum of which could be 12 . Reflective scores were assessed from the hour since the last dose of study medication.
Time Frame: 14 days minus baseline
Population: The analysis was per protocol. 15 patients were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCl Nasal Spray, 0.6% | Azelastine HCl Nasal Spray, 0.1%
Number analyzed (Participants) | 67 | 68
Units on a scale | 4.28 (2.63) | 4.15 (2.63)

2. Primary Outcome: Mean Change in Reflective Total Ocular Symptom Scores (rTOSS) From Baseline
Description: Responses to patient-completed diaries for reflective Total Ocular Symptom Scores (rTOSS). TOSS is composed of 3 individual assessments of ocular symptoms (itching/burning, tearing/watering, redness) each of the 3 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 3 assessments are then added together for a composite score (TOSS score), the maximum of which could be 9 . Reflective scores were assessed from the hour since the last dose of study medication.
Time Frame: 14 days minus baseline
Population: The analysis was per protocol. 15 patients were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCl Nasal Spray, 0.6% | Azelastine HCl Nasal Spray, 0.1%
Number analyzed (Participants) | 67 | 68
Units on a scale | 4.22 (2.69) | 4.04 (2.45)

3. Primary Outcome: Mean Change in Instantaneous Total Nasal Symptom Scores (iTNSS) From Baseline
Description: Responses to patient-completed diaries for instantaneous Total Nasal Symptom Scores (iTNSS). TNSS is composed of 4 individual assessments, which included runny nose, itchy nose, stuffy nose, and sneezing; each of the 4 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 4 assessments are then added together for a composite score (TNSS score), the maximum of which could be 12 . Instantaneous scores were assessed at the time of daily dosing.
Time Frame: 14 days minus baseline
Population: The analysis was per protocol. 15 patients were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCl Nasal Spray, 0.6% | Azelastine HCl Nasal Spray, 0.1%
Number analyzed (Participants) | 67 | 68
Units on a scale | 2.64 (2.13) | 2.49 (2.07)

4. Primary Outcome: Mean Change in Instantaneous Total Ocular Symptom Scores (iTOSS) From Baseline
Description: Responses to patient-completed diaries for instantaneous Total Ocular Symptom Scores (iTOSS). TOSS is composed of 3 individual assessments of ocular symptoms (itching/burning, tearing/watering, redness) each of the 3 assessments were rated using a 4 point scale that ranged in whole units from 0 (none) to 3 (severe). All 3 assessments are then added together for a composite score (TOSS score), the maximum of which could be 9 . Instantaneous scores were assessed at the time of daily dosing.
Time Frame: 14 days minus baseline
Population: The analysis was per protocol. 15 patients were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Olopatadine HCl Nasal Spray, 0.6% | Azelastine HCl Nasal Spray, 0.1%
Number analyzed (Participants) | 67 | 68
Units on a scale | 2.76 (2.21) | 2.54 (2.08)

ADVERSE EVENTS:
Arm/Group | Olopatadine HCl Nasal Spray, 0.6% | Azelastine HCl Nasal Spray, 0.1%
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No